CLINICAL TRIAL: NCT03779022
Title: MicroRNA and Relevant Biomarkers of Breast Cancer in Patients Undergoing Neoadjuvant Treatment
Brief Title: miRNA and Relevant Biomarkers of BC Patients Undergoing Neoadjuvant Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cui Yimin (Other)
Responsible Party: Sponsor-Investigator, Cui Yimin, Director of pharmacy, M.D & Ph.D, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Other Study IDs: miRNA-NAT-BC
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; biomarker; neoadjuvant treatment; microRNA; response
MeSH Terms: conditions — Breast Neoplasms | interventions — MicroRNAs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For each patient, 4 mL of peripheral blood will be collected as per predesigned schedule. Within 4 hours of blood drawl, samples will be centrifuged at 1500g for 10min at 4℃ to separate the plasma supernatant. The plasma and the blood cell will be aliquoted and stored at -80℃ until analysis, respectively.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sensitive: Sensitive group was defined ad complete response (CR) and/or partial response (PR). Blood samples for microRNA were collected before neoadjuvant chemotherapy, evaluation of clinical disease response and surgery.
  Interventions: Genetic: microRNA
- Resistant: Resistant group was defined ad progression disease (PD) and/or stable disease (SD). Blood samples for microRNA were collected before neoadjuvant chemotherapy, evaluation of clinical disease response and surgery.
  Interventions: Genetic: microRNA

INTERVENTIONS:
Genetic: microRNA — The level of microRNA in plasma will be detected by TaqMan in screening phase and by quantitative Real-time PCR (qRT-PCR) in validation phase.

SUMMARY:
MicroRNA (miRNA) is a type of endogenous non-coding RNA. They are responsible for post-transcriptional regulation and participate in many vital biological processes. Expression profiling has shown that miRNAs can distinguish between normal breast and tumor tissues. In recent years, circulating miRNAs have become promising biomarkers based on their stability and their non-invasive testing and feasibility in clinical practices.

DETAILED DESCRIPTION:
Current reports showed that serum microRNA expression could be used as an early marker for determining the breast cancer risk. The concentrations of some circulating microRNAs in human breast cancer have been correlated with tumor development and progression. Aberrant miRNA expression may be involved in drug resistance to various chemotherapeutic agents in breast cancer. Therefore, we hope to investigate the value of miRNAs in predicting the effect in breast cancer neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Early breast cancer patients;
2. Stage II-III disease;
3. sign informed consent form;
4. receive neoadjuvant treatment;
5. Age between 18-75.

Exclusion Criteria:

1. Women during pregnancy;
2. Metastasis patients or stage IV breast cancer patients;
3. Male breast cancer patients;
4. Inflammatory breast cancer patients;
5. Patients with neoadjuvant endocrine treatment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients was eligible.
Study Population: Female, Breast Cancer, >18 years,<75 years, early stage breast cancer patients, with Stage II-III disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-11-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response | Every 2 cycles, up to surgery (each cycle is 21 days)
  Clinical disease response was evaluated for every two cycles of chemotherapy till surgery with RECIST criteria (RECIST 1.1). Resistant group was defined ad progression disease (PD) and/or stable disease (SD).Evaluation in breast lesions by MRI or mammography. The same imaging methods were used throughout treatment for a given patient. Blood samples for microRNA were collected before neoadjuvant chemotherapy, evaluation of clinical disease response and surgery.
  Clinical disease response was evaluated for every two cycles of chemotherapy till surgery with RECIST criteria (RECIST 1.1). Evaluation in breast lesions by MRI or mammography. The same imaging methods were used throughout treatment for a given patient.

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Cui, Ph.D & M.D, Study Director — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
We would not like to share individual participant data (IPD) but share the result after statistical analysis. If IPD was needed, please contact us by e-mail.

REFERENCES:
- [Background] Li Q, Liu M, Ma F, Luo Y, Cai R, Wang L, Xu N, Xu B. Circulating miR-19a and miR-205 in serum may predict the sensitivity of luminal A subtype of breast cancer patients to neoadjuvant chemotherapy with epirubicin plus paclitaxel. PLoS One. 2014 Aug 19;9(8):e104870. doi: 10.1371/journal.pone.0104870. eCollection 2014. PMID 25137071
- [Background] Wang H, Tan G, Dong L, Cheng L, Li K, Wang Z, Luo H. Circulating MiR-125b as a marker predicting chemoresistance in breast cancer. PLoS One. 2012;7(4):e34210. doi: 10.1371/journal.pone.0034210. Epub 2012 Apr 16. PMID 22523546
- [Background] Zhao R, Wu J, Jia W, Gong C, Yu F, Ren Z, Chen K, He J, Su F. Plasma miR-221 as a predictive biomarker for chemoresistance in breast cancer patients who previously received neoadjuvant chemotherapy. Onkologie. 2011;34(12):675-80. doi: 10.1159/000334552. Epub 2011 Nov 23. PMID 22156446
- [Background] Zhu W, Liu M, Fan Y, Ma F, Xu N, Xu B. Dynamics of circulating microRNAs as a novel indicator of clinical response to neoadjuvant chemotherapy in breast cancer. Cancer Med. 2018 Sep;7(9):4420-4433. doi: 10.1002/cam4.1723. Epub 2018 Aug 11. PMID 30099860